CLINICAL TRIAL: NCT01677559
Title: Phase I Study Combining MLN8237 With Nab-Paclitaxel in Patients With Advanced Solid Malignancies
Brief Title: Combining MLN8237 With Nab-Paclitaxel in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201210123
Record Dates: First submitted 2012-08-27; First posted 2012-09-03 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Adenocarcinoma; Pancreatic Neoplasms
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms | interventions — MLN 8237; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level 0 (Experimental): MLN8237 20 mg BID Days 1, 2 and 3 of each week for 3 weeks out of a 4 week cycle.
  nab-Paclitaxel 100 mg/m2 IV Day 1 of each week for 3 weeks out of a 4 week cycle.
  Interventions: Drug: MLN8237; Drug: nab-Paclitaxel
- Dose Level 1 (Experimental): MLN8237 30 mg BID Days 1, 2 and 3 of each week for 3 weeks out of a 4 week cycle.
  nab-Paclitaxel 100 mg/m2 IV Day 1 of each week for 3 weeks out of a 4 week cycle.
  Interventions: Drug: MLN8237; Drug: nab-Paclitaxel
- Dose Level 2 (Experimental): MLN8237 40 mg BID Days 1, 2 and 3 of each week for 3 weeks out of a 4 week cycle.
  nab-Paclitaxel 100 mg/m2 IV Day 1 of each week for 3 weeks out of a 4 week cycle.
  Interventions: Drug: MLN8237; Drug: nab-Paclitaxel
- Dose Level 3 (Experimental): MLN8237 50 mg BID Days 1, 2 and 3 of each week for 3 weeks out of a 4 week cycle.
  nab-Paclitaxel 100 mg/m2 IV Day 1 of each week for 3 weeks out of a 4 week cycle.
  Interventions: Drug: MLN8237; Drug: nab-Paclitaxel
- MTD Expansion Phase (Experimental): MLN8237 as determined during the dose escalation phase on Days 1, 2 and 3 of each week for 3 weeks out of a 4 week cycle.
  nab-Paclitaxel 100 mg/m2 IV Day 1 of each week for 3 weeks out of a 4 week cycle.
  Interventions: Drug: MLN8237; Drug: nab-Paclitaxel

INTERVENTIONS:
Drug: MLN8237
Drug: nab-Paclitaxel
  Other Names: Abraxane; Coroxane; Capxol

SUMMARY:
This phase I trial studies the side effects and the best dose of MLN8237 (alisertib) when given together with paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel) in treating patients with solid malignancies that are metastatic or cannot be removed by surgery. Alisertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as nab-paclitaxel work by killing the cells or by stopping them from dividing. Giving alisertib together with nab-paclitaxel may provide a more effective anticancer treatment with fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures to not exist or are no longer effective (dose-escalation cohorts only).
* Patient must have a histologically or cytologically confirmed diagnosis of pancreatic cancer or poorly differentiated neuroendocrine tumor and must have been treated with a regimen with known benefit for pancreatic cancer or poorly differentiated neuroendocrine tumor (MTD expansion cohort only).
* Patient must have measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Patient must have disease that is easily accessible for a core biopsy as determined by the treating physician or study PI. Patient must agree to the mandatory biopsies at baseline and end of Cycle 2 (MTD expansion cohort only, and at the discretion of the PI/PI optional).
* Patient must be ≥ 18 years of age.
* Patient must have an ECOG performance status of 0 or 1
* Patient must have normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin > 9.0 g/dL
  * Total bilirubin ≤ institutional ULN
  * AST and ALT < 1.5 x ULN (or < 5 x ULN if known liver metastases)
  * Calculated creatinine clearance must be > 40 mL/min (by Cockcroft-Gault)
* If a female of childbearing potential (defined as a female who is non-menopausal or surgically sterilized), patient must be willing to use an acceptable method of birth control (i.e., hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. If a male with a partner who is a female of childbearing potential, patient must agree to use an acceptable method of contraception during the entire study treatment period through 4 months after the last dose of MLN8237. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patient must be able to take oral medication and to maintain a fast as required for 2 hours before and 1 hour after MLN8237 administration.
* Patient (or legally authorized representative if applicable) must be able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Patient must not have received chemotherapy or radiotherapy ≤ 4 weeks or 5 half-lives prior to study entry.
* Patient must not have had radiation therapy to more than 25% of the bone marrow. Whole pelvic radiation is considered to be over 25%.
* Patient must not have a history of other malignancy ≤ 2 years previous with the exception of basal cell or squamous cell carcinoma of the skin which was treated with local resection only, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Patient must not have had a prior allogeneic bone marrow or organ transplantation.
* Patient must not have previously received nab-paclitaxel.
* Patient must not have received any other investigational agents within 14 days prior to study enrollment.
* Patient must not have known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to either MLN8237 or nab-paclitaxel, or other agents used in the study.
* Patient must not have been treated with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine, or Phenobarbital, or rifampin, rifabutin, rifapentine, or St. John's wort within 14 days prior to the first dose of MLN8237.
* Patient must not have received any previous treatment with any Aurora-kinase inhibitors (MTD expansion cohort only).
* Patient must not have a history of gastric resection (MTD expansion cohort only).
* Patient must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient must not have ≥ grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient must not have a known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease.
* Patient must not have a requirement for supplemental oxygen.
* Patient must not require constant administration of a proton pump inhibitor, H2 antagonist, or pancreatic enzymes. Intermittent uses of antacids or H2 antagonists are allowed.
* Patient must not have QTc > 500ms within 14 days before enrollment.
* Patient must not have had a myocardial infarction within 6 months prior to enrollment or have New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patient must not be pregnant and/or breastfeeding.
* Patient must not be known to be HIV-positive on combination antiretroviral because of the potential for pharmacokinetic interactions with MLN8237 or Abraxane. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Inclusion of Women and Minorities

Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-05-07 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Completion of cycle 1
Dose-limiting toxicities (DLTs) | Completion of cycle 1
  Hematologic DLT is defined as any of the following that occurs during the first cycle that is attributed as possibly, probably or definitely related to the study treatment:
  * Grade 4 neutropenia > 7 days duration
  * Febrile neutropenia of any duration with temperature ≥ 38.5 °C
  * Grade 4 thrombocytopenia > 7 days duration
  Non-hematologic DLT is defined as any possibly, probably, or definitely related grade 3 or grade 4 non-hematologic toxicity that occurs during the first cycle with the following specific exceptions:
  * Grade 3 fatigue
  * Grade 3 or 4 nausea, vomiting, or anorexia that returns to Grade 1 prior to the start of Cycle 2
  * Grade 3 non-hematological laboratory abnormalities that resolve to grade 1 or baseline prior to the start of Cycle 2
  Any delay in treatment >14 days that is possibly, probably, or definitely related to study treatment will be considered a DLT.

SECONDARY OUTCOMES:
Antitumor activity of MLN8237 and nab-paclitaxel combination therapy | 60 days
  Overall response rate (ORR = CR + PR) as a preliminary measure

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Wang-Gillam, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim KH, Opyrchal M, Acharya A, Boice N, Wu N, Gao F, Webster J, Lockhart AC, Waqar SN, Govindan R, Morgensztern D, Picus J, Tan BR, Baggstrom MQ, Maher CA, Wang-Gillam A. Phase 1 study combining alisertib with nab-paclitaxel in patients with advanced solid malignancies. Eur J Cancer. 2021 Sep;154:102-110. doi: 10.1016/j.ejca.2021.06.012. Epub 2021 Jul 10. PMID 34256279
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu